CLINICAL TRIAL: NCT00818571
Title: An Open-label, Parallel Group Study to Determine the PK of 25 and 50 mg OD Single and Multiple Dose Over 14 Days, of Vildagliptin and Its Metabolites in Renal Impaired Patients Compared to Matching Healthy Volunteers
Brief Title: Pharmacokinetics of Vildagliptin in Mild, Moderate and Severe Renal Impaired Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237B2202; 2008-004565-25 (EudraCT Number)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-01

CONDITIONS: Renal Impairment; Diabetes
Keywords: Renal impairment; Diabetes; vildagliptin; Galvus; Eucreas
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus | interventions — Vildagliptin

ARMS (4):
- Vildagliptin 25 mg qd in Renal Impaired (RI) patients (Experimental)
  Interventions: Drug: Vildagliptin
- Vildagliptin 50 mg qd in RI Patients (Experimental)
  Interventions: Drug: Vildagliptin
- Vildagliptin 25 mg qd in matched Healthy Volunteer (HV) (Experimental)
  Interventions: Drug: Vildagliptin
- Vildagliptin 50 mg qd in matched HV (Experimental)
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Mild, moderate and severe renal impaired patients receiving 25 mg vildagliptin once daily
  Arms: Vildagliptin 25 mg qd in Renal Impaired (RI) patients
Drug: Vildagliptin — Mild, moderate and severe renal impaired patients receiving 50 mg vildagliptin once daily
  Arms: Vildagliptin 50 mg qd in RI Patients
Drug: Vildagliptin — Matching healthy volunteers receiving 25 mg vildagliptin once daily.
  Arms: Vildagliptin 25 mg qd in matched Healthy Volunteer (HV)
Drug: Vildagliptin — Matching healthy volunteers receiving 50 mg vildagliptin once daily
  Arms: Vildagliptin 50 mg qd in matched HV

SUMMARY:
This study assess the pharmacokinetics of vildagliptin in mild, moderate and severe renal impaired patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild (CrCl from 50 to ≤80 ml/min), moderate (CrCl from 30 to <50 ml/min) and severe (CrCl of <30 ml/min) renal function, preferably type 2 diabetic and matching healthy volunteers CrCl of >80 ml/min

Exclusion Criteria:

* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, acute metabolic diabetic complications, treatment of a DPP-4 inhibitor 30 days prior to baseline, renal transplant history

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Measure: pharmacokinetics of vildagliptin and its metabolites | 14 days

SECONDARY OUTCOMES:
Measure: safety assessments will include vital signs, electrocardiograms and adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigator Site, Moscow, Russia

REFERENCES:
- See also: Results for CLAF237B2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2949